CLINICAL TRIAL: NCT02107612
Title: Development of Minimally Invasive Splinted Dental Implants to Stabilize Mandibular Overdentures, a Randomized Clinical Trial
Brief Title: Randomized Study For Minimally Invasive Splinted Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Concepcion, Chile (Other)
Collaborators: Public Health Service of Chile (Unknown)
Responsible Party: Principal Investigator, Jorge Jofre, Jorge Jofre DDs, PhD, University of Concepcion, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FONDEF V09E0007
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Jaw, Edentulous
Keywords: Mini-Dental Implant; Implant-Supported Dental Prosthesis; Minimally Invasive Surgical procedures; Overdentures; Aged
MeSH Terms: conditions — Jaw, Edentulous | interventions — Dental Implants; Dentures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Integrated system to insert two splinted (bar) miniimplants (Experimental): Participants were randomly assigned to experimental group following a simple randomization procedure (computer-generated list of random numbers). Allocation by telephone was carried out with an independent collaborator.
  Interventions: Device: Integrated system to insert two splinted (bar) mini dental implants for mandibular overdenture
- Denture (Active Comparator): Participants were randomly assigned to comparator group following a simple randomization procedure (computer-generated list of random numbers). Allocation by telephone was carried out with an independent collaborator.
  Interventions: Other: Denture

INTERVENTIONS:
Device: Integrated system to insert two splinted (bar) mini dental implants for mandibular overdenture
  Other Names: Easy2Fix
  Arms: Integrated system to insert two splinted (bar) miniimplants
Other: Denture
  Arms: Denture

SUMMARY:
The purpose of this study was to evaluate the effect of a integrated system for inserting two splinted minimally-invasive implants, to retain mandibular over dentures, on the quality of life of edentulous patients.

ELIGIBILITY:
Inclusion Criteria:

* Edentulous
* Men and women
* Between 45 and 90 years of age
* Who had a persistent loss of stability and retention of their conventional mandibular dentures
* Without temporomandibular disorders

Exclusion Criteria:

* Uncontrolled systemic disease (eg, hypertension, diabetes)
* Severe osteoporosis (bone mineral density > 2.5 SD below the young adult reference mean, plus 1 or more fragility fractures) and/or taking bisphosphonates
* Mental disorders
* Who had received radiotherapy in the 18 months prior to the trial

Ages: 45 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2004-07; Primary Completion 2006-04 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | One year
  Quality of life was assessed using the Oral Health Impact Profile (OHIP) for assessing health-related quality of life in edentulous adults (EDENT) scale with 19 items.

SECONDARY OUTCOMES:
Incidence of complications | Two years
  Complications: infection, implant failure, presence of signs and symptoms of peri-implant mucositis.

OTHER OUTCOMES:
Average marginal bone loss in the peri-implant zone | Two years
Average of maximal bite force | Fifteen months
Mini-implant survival rate | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Jofre, DDS, PhD, Principal Investigator — University of Concepcion
Locations (1):
- University of Concepción, Concepción, Región Del Bio Bio, Chile

REFERENCES:
- [Result] Jofre J, Castiglioni X, Lobos CA. Influence of minimally invasive implant-retained overdenture on patients' quality of life: a randomized clinical trial. Clin Oral Implants Res. 2013 Oct;24(10):1173-7. doi: 10.1111/j.1600-0501.2012.02529.x. Epub 2012 Jul 4. PMID 22762359
- [Result] Jofre J, Cendoya P, Munoz P. Effect of splinting mini-implants on marginal bone loss: a biomechanical model and clinical randomized study with mandibular overdentures. Int J Oral Maxillofac Implants. 2010 Nov-Dec;25(6):1137-44. PMID 21197490
- [Result] Jofre J, Conrady Y, Carrasco C. Survival of splinted mini-implants after contamination with stainless steel. Int J Oral Maxillofac Implants. 2010 Mar-Apr;25(2):351-6. PMID 20369095
- [Result] Jofre J, Hamada T, Nishimura M, Klattenhoff C. The effect of maximum bite force on marginal bone loss of mini-implants supporting a mandibular overdenture: a randomized controlled trial. Clin Oral Implants Res. 2010 Feb;21(2):243-9. doi: 10.1111/j.1600-0501.2009.01834.x. PMID 20070758